CLINICAL TRIAL: NCT04277351
Title: Role of Auditory Cortical Oscillations in Speech Processing and Its Dysfunction in Dyslexia Through Transcranial Alternating Current Stimulation
Brief Title: Role of Auditory Cortical Oscillations in Speech Processing and Dyslexia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Geneva, Switzerland (Other)
Collaborators: Wyss Center for Bio and Neuroengineering (Other)
Responsible Party: Principal Investigator, Anne-Lise Giraud, Professor, University of Geneva, Switzerland
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: PHONOSTIM
Record Dates: First submitted 2020-02-13; First posted 2020-02-20 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Dyslexia
MeSH Terms: conditions — Dyslexia | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant
Masking Description: One of three different tACS conditions is administered to all participant during three experimental days. The conditions differ in the frequency of stimulation (condition 1 and 2) and in whether the stimulation is active or faked (sham). The order of the three stimulation conditions is counterbalanced across participants, who are not aware of which tACS condition they are undergoing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- tACS in individuals with and without dyslexia (Experimental): Each participant in both the group of normo-readers and individuals with dyslexia receive all tACS stimulation conditions (fixed frequencies and sham) over different experimental days.
  Interventions: Device: Transcranial alternating current stimulation

INTERVENTIONS:
Device: Transcranial alternating current stimulation — Focal transcranial stimulation over auditory cortex by means of 5 electrodes delivering an electric current (max. 2mA). In addition to active stimulation, also a placebo (sham) stimulation is employed as a control condition. All subjects included in the study receive all tACS stimulation conditions.

SUMMARY:
This study aims at investigating the role of low-gamma activity in phonemic encoding and its implication in dyslexia. Indeed, a phonological deficit, i.e. a difficulty in perceiving the sounds of speech, is strongly suspected in dyslexia but has never been conclusively associated with a specific underlying mechanism.

The study employs transcranial alternating current stimulation in adults with and without dyslexia to exploit the effect of the stimulation on phonemic processing and neural activity measured with electroencephalography. In doing so, it would be possible to establishing a causal link between gamma oscillations and the phonological deficit in dyslexia.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old;
* French native speakers;
* normally-hearing;
* intellectual quotient (IQ) around average;
* for the dyslexia group: previous diagnosis of dyslexia as assessed by a speech therapist.

Exclusion Criteria:

* Presence of metal or electronic implants in the brain/skull;
* Presence of metal or electronic device at other in other parts of the body;
* Have experienced a seizure or a loss of consciousness or a severe head trauma;
* Severe brain related illness ;
* Intake of central nervous system-effective medication;
* Pregnant and nursing women;
* Relatives affected by epilepsy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Measure low-gamma neural oscillations with electroencephalography recordings | 6 hour
  Auditory-steady state responses to auditory stimuli are measured to assess specific differences between individuals with dyslexia and normo-readers, and between the different tACS stimulation conditions before, after and 1h after the 20 min. tACS stimulation.
  These neural correlated are estimated by considering the power of EEG signal at the frequency used to modulate the auditory stimuli.
Changes in linguistic performance through a battery of behavioral tests | 6 hours
  Measurement of phonemic and syllabic processing (pseudoword repetition and spoonerism test), and reading (reading a 3 min. text, both accuracy and reading speed are considered) skills. These tests are repeated before, after and 1h after the tACS stimulation.

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Lise Giraud, Prof., Principal Investigator — University of Geneva
Locations (1):
- Campus Biotech Geneva, Geneva, Switzerland

REFERENCES:
- [Background] Lehongre K, Ramus F, Villiermet N, Schwartz D, Giraud AL. Altered low-gamma sampling in auditory cortex accounts for the three main facets of dyslexia. Neuron. 2011 Dec 22;72(6):1080-90. doi: 10.1016/j.neuron.2011.11.002. PMID 22196341